CLINICAL TRIAL: NCT07251751
Title: Forward Versus Backward Gait Training on Functional Abilities in Children With Spastic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ramy Abdulmoneem Abdullah Khidr, Principal Investigator and Physiotherapist, Ministry of Health - Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ramy Gait training in C.P
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Spastic Cerebral Palsy
Keywords: Gait Training
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (designed physical therapy program) (Active Comparator): participants will receive designed physical therapy exercises only
  Interventions: Behavioral: control group ( designed physical therapy program)
- forward gait training (Experimental): participants will receive designed physical therapy exercises beside forward gait training.
  Interventions: Behavioral: forward gait training
- backward gait training (Experimental): participants will receive designed physical therapy exercises beside backward gait training.
  Interventions: Behavioral: backward gait training

INTERVENTIONS:
Behavioral: control group ( designed physical therapy program) — Participants receive traditional physical therapy exercises focusing on stretching, strengthening, and balance training for the same duration as the experimental groups.
  Arms: control group (designed physical therapy program)
Behavioral: forward gait training — The training program consists of forward walking exercises conducted three times per week for three successive months under the supervision of a physical therapist.
  Arms: forward gait training
Behavioral: backward gait training — The training program consists of backward walking exercises conducted three times per week for three successive months under the supervision of a physical therapist.
  Arms: backward gait training

SUMMARY:
This study aims to compare the effects of forward versus backward gait training on functional abilities in children with spastic cerebral palsy. Participants will receive gait training sessions focusing on either forward or backward walking to evaluate improvements in balance, mobility, and gross motor function.

DETAILED DESCRIPTION:
> Cerebral palsy is a common neurological disorder in children that affects movement and posture. Spastic cerebral palsy is characterized by muscle stiffness and impaired motor control, which limits the child's functional mobility.

Gait training is an essential part of rehabilitation programs for children with cerebral palsy. Previous studies have shown that both forward and backward walking can improve motor performance, but limited evidence exists comparing the two methods directly.

The present randomized clinical trial aims to compare the effects of forward gait training versus backward gait training on functional abilities in children with spastic cerebral palsy. Participants will be randomly assigned into three groups: group (A) will receive a designed physical therapy program. group (B) will receive the same program with forward gait training on treadmill. group (C) will receive the same designed physical therapy program beside backward gait training on treadmill three times weekly over three successive months.

Outcome measures will include muscle strength of measurements, range of motion of lower limb,gait pattern changes and gross motor function measurements.

ELIGIBILITY:
Inclusion Criteria:1-All children will be spastic diplegic cerebral palsy. 2- Age will be ranged from 6-9 years old. 3. They will have spasticity grade 1 to 1+ according to Modified Ashwarth's Scale (Appendix II).

4. Both genders will be included. 5. Their gross motor function ability will be selected at level I, II according to Gross Motor Function Classification System (GMFCS).

6. They will be able to understand and follow verbal commands included in evaluation and training.

Exclusion Criteria:

1- Any surgical intervention in upper or lower limbs. 2¬- Any type of fracture. 3- Visual and/or auditory defects. 4- Other neurological conditions rather than CP. 5- Significant tightness or fixed deformity of lower limbs and spine. 6- Congenital heart disease.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-88) score | Baseline and after three months of intervention
  The GMFM-88 will be used to assess changes in gross motor function in children with spastic cerebral palsy before and after the intervention. Higher scores indicate better motor performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ramy A Khidr, PhD, Principal Investigator — El shohadaa Central Hospital
Locations (1):
- El Shohadaa Central Hospital, Shibīn al Kawm, Monoufia, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is conducted locally for academic and clinical purposes only.

REFERENCES:
- [Background] Keep H, Luu L, Berson A, Garland SJ. Validity of the Handheld Dynamometer Compared with an Isokinetic Dynamometer in Measuring Peak Hip Extension Strength. Physiother Can. 2016;68(1):15-22. doi: 10.3138/ptc.2014-62. PMID 27504043